CLINICAL TRIAL: NCT00742716
Title: An Open Label, Four Week, Dose Escalating Pharmacokinetic, Pharmacodynamic, Efficacy and Safety Study of CTA018 Injection in Subjects With Stage 5 Chronic Kidney Disease With Secondary Hyperparathyroidism on Hemodialysis
Brief Title: Safety Study of CTA018 Injection to Treat Stage 5 Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO IP Holdings II, Inc. (Industry)
Responsible Party: Sponsor
Organization: OPKO Health, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTA018-CL-2002
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism; Chronic Renal Insufficiency; Chronic Renal Failure
Keywords: Parathyroid Diseases; Renal Insufficiency; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D; Hyperparathyroidism; Renal Insufficiency, Chronic; Kidney Diseases; Kidney Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary; Kidney Failure, Chronic; Parathyroid Diseases; Renal Insufficiency; Hyperparathyroidism; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CTA018 Injection low dose (Experimental): Low dose IV 3 times a week for 4 weeks
  Interventions: Drug: CTA018 Injection
- CTA018 Injection low to mid dose (Experimental): low to mid dose IV 3 times a week for 4 weeks
  Interventions: Drug: CTA018 Injection
- CTA018 Injection mid to high dose (Experimental): mid to high dose IV 3 times a week for 4 weeks
  Interventions: Drug: CTA018 Injection
- CTA018 Injection high dose (Experimental): high dose IV 3 times a week for 4 weeks
  Interventions: Drug: CTA018 Injection

INTERVENTIONS:
Drug: CTA018 Injection — Comparison of different dosages of drug

SUMMARY:
This study will investigate the levels of CTA018 in the body over time (pharmacokinetics, PK) in patients with chronic kidney disease (CKD) and secondary hyperparathyroidism (SHPT), undergoing regular hemodialysis. This study will also investigate the safety and effects of different strengths of CTA018, on parathyroid hormone (PTH) levels.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 35
* On maintenance hemodialysis three times per week
* Serum iPTH value greater than or equal to 300 pg/mL and lower than or equal to 1000 pg/mL
* Adjusted or total serum calcium value greater than or equal to 8.4 mg/dL and lower than 10.0 mg/dL
* Serum phosphorus value greater than or equal to 2.5 mg/dL and lower than or equal to 5.5 mg/dL
* Serum 25-hydroxyvitamin D level greater than or equal to 15 ng/mL
* Willing and able to discontinue vitamin D and/or bone metabolism therapy for at least 2 weeks prior to administration of Study Drug, and the length of study

Exclusion Criteria:

* On bisphosphonates for at least three months prior to first dose of Study Drug
* Currently taking cytochrome P450 3A inhibitors and/or inducers
* Abnormal liver functions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To assess the single and repeat dose pharmacokinetics (PK) of CTA018 Injection | Day 1 and 12 of each dose level
To investigate the safety of CTA018 Injection | Throughout the study

SECONDARY OUTCOMES:
To investigate the pharmacodynamic (PD) intact parathyroid hormone (iPTH) response following CTA08 Injection | Throughout the study
To determine the efficacy of CTA018 Injection to reduce serum iPTH | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Joel Melnick, MD, Study Director — OPKO Renal
Locations (12):
- United States (5):
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Western New England Renal & Transplant Associates (WNERTA), Springfield, Massachusetts
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - U.S. Renal Care, Fort Worth, Texas
- Canada (7):
  - Capital District Heatlth Authority: Centre for Clinical Research, Halifax, Nova Scotia
  - St. Joseph's Health Care London, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Hôpital Charles-Lemoyne, Greenfield Park, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Hospital de Verdun, Verdun, Quebec